CLINICAL TRIAL: NCT01696643
Title: Phase 3 Study to Evaluate the Long-Term Safety and Tolerability of CB-5945 for the Treatment of Opioid-Induced Constipation in Adults Taking Opioid Therapy for Chronic Non-Cancer Pain
Brief Title: Safety Study of CB-5945 for the Treatment of Opioid-Induced Constipation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A review of blinded data indicates that the number of participant exposures needed to reach ICH standards has been met
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2402-006; 5945-SOIC-12-05 (Other: Cubist Study Number)
Record Dates: First submitted 2012-09-21; First posted 2012-10-01 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Opioid-Induced Constipation
Keywords: Opioid; Constipation; Chronic; Pain
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- CB-5945 (Experimental): 0.25 milligrams (mg) CB-5945, administered orally, twice daily (BID) for 52 weeks
  Interventions: Drug: CB-5945
- Placebo (Placebo Comparator): Placebo, administered orally, BID for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CB-5945
  Other Names: Bevenopran
  Arms: CB-5945
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of CB-5945 for the treatment of opioid-induced constipation (OIC) in adults taking opioid therapy for chronic non-cancer pain.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, placebo-controlled, parallel-group study in participants with OIC taking opioid therapy for chronic non-cancer pain. Approximately 1,400 participants (approximately 700 participants per treatment group) with OIC will be randomized at approximately 225 study centers to receive either 0.25 milligrams (mg) CB-5945 twice daily (BID) or a matching placebo BID for the 52-week double-blind treatment period, followed by a 4-week follow-up period. All randomized participants will be evaluated for safety, tolerability, and quality of life from the first dose of study drug through Week 56.

ELIGIBILITY:
Inclusion Criteria:

* Is taking a stable daily dose of opioids of ≥30-mg morphine-equivalent total daily dose (METDD) for chronic non-cancer pain
* Has constipation that is caused by the chronic use of opioids
* Is willing to use only the study-provided laxative(s) and to discontinue use of all other laxatives, enemas, stool softeners, and other medications to treat constipation (for example, lubiprostone) during the study period (from Screening until the last study assessment).
* Is able and willing to refrain from facilitating defecation via manual maneuvers (for example, digital evacuation or support of the pelvic floor) during the study period (from Screening to the last study assessment)

Exclusion Criteria:

* Has gastrointestinal (GI) or pelvic disorders known to affect bowel transit (for example, obstruction) or contribute to bowel dysfunction
* Has evidence of intestinal obstruction
* Has a history of rectal bleeding not due to hemorrhoids or fissures
* Has an active malignancy of any type (participants with a history of successfully treated malignancy >5 years before the scheduled administration of study medication and participants with treated basal or squamous cell cancer may be enrolled)
* Is taking antispasmodics (for example, dicyclomine), antidiarrheals (for example, loperamide), prokinetics (for example, metoclopramide), or locally acting chloride channel activators (for example, lubiprostone)
* Is taking non-opioid medications known to cause constipation (for example, iron sulfate therapy or tricyclic antidepressants)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1407 (Actual)
Dates: Start 2012-10-12 (Actual); Primary Completion 2014-07-21 (Actual); Study Completion 2014-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CB-5945 | Placebo
Started | 703 | 704
Received at Least 1 Dose of Study Drug | 701 | 702 (2 participants randomized to placebo took CB-5945. Their results are included in the CB-5945 group.)
Completed | 174 | 169
Not Completed | 529 | 535
Not completed — Adverse Event | 15 | 7
Not completed — Death | 1 | 2
Not completed — Lack of Efficacy | 3 | 0
Not completed — Lost to Follow-up | 67 | 67
Not completed — Physician Decision | 3 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 7 | 7
Not completed — Study Terminated by Sponsor | 286 | 294
Not completed — Withdrawal by Subject | 142 | 149
Not completed — Participant on Restricted Bed Rest | 1 | 0
Not completed — Site Error | 2 | 1
Not completed — Participant Incarcerated | 0 | 1
Not completed — Medical Monitor Decision | 0 | 2
Not completed — Participant Did Not Receive Study Drug | 2 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug. Two participants were randomized to the Placebo Arm but were administered CB-5945 instead. As a result, these 2 participants were included in the CB-5945 Arm for analysis.
Groups:
- CB-5945: 0.25 mg CB-5945, administered orally, BID for 52 weeks
- Total: Total of all reporting groups
Arm/Group | CB-5945 | Placebo | Total
Number analyzed (Participants) | 703 | 700 | 1403
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.00) | 53.9 (10.21) | 54.2 (10.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 437 | 417 | 854
  Male | 266 | 283 | 549
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 41 | 60
  Not Hispanic or Latino | 676 | 649 | 1325
  Unknown or Not Reported | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 4 | 11
  Asian | 11 | 11 | 22
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 117 | 122 | 239
  White | 563 | 555 | 1118
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 26 | 28 | 54
  United States | 677 | 672 | 1349

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as any adverse event (AE) that occurred from the time of first dose of the study drug through the last study evaluation or pre-existing AEs that were aggravated in severity or frequency during the dosing period. The percentages of participants with at least 1 TEAE, with at least 1 drug-related TEAE (drug-related included "possibly related" or "related" as deemed by the Investigator; it also included events if causality was missing), and who discontinued from treatment due to a TEAE are presented. A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through Week 56
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | CB-5945 | Placebo
Number analyzed (Participants) | 703 | 700
percentage of participants
  Had at least 1 TEAE | 58.5 | 54.0
  Had at least 1 drug-related TEAE | 19.9 | 12.1
  Discontinued treatment due to a TEAE | 10.0 | 5.7

2. Secondary Outcome: Change From Baseline in Mean Daily Opioid Dose at Weeks 49-52
Description: Throughout the study, participants were asked to record changes in maintenance opioid consumption and use of opioid analgesics for breakthrough or exacerbation of pain in a paper diary. Opioid consumption (including rescue opioids) of each participant was converted to an oral morphine-equivalent total daily dose (METDD). Opioid consumption (in milligrams of METDD) was summarized in 4-week intervals. The change from baseline to Weeks 49-52 is summarized.
Time Frame: Baseline, Weeks 49-52
Population: All randomized participants who received at least 1 dose of study drug and had evaluable METDD data. Two participants were randomized to the Placebo Arm but were administered CB-5945 instead. As a result, these 2 participants were included in the CB-5945 Arm for analysis.
Measure: Mean (Standard Deviation); unit: milligrams of METDD
Arm/Group | CB-5945 | Placebo
Number analyzed (Participants) | 672 | 664
milligrams of METDD | -12.456 (90.2190) | -12.297 (88.8681)

3. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation-Quality of Life (PAC-QOL) Questionnaire at Week 52
Description: The PAC-QOL questionnaire contains a total of 28 items, each rated within 4 subscales: physical discomfort, psychosocial discomfort, worries and concerns, and satisfaction. Each item was rated on a 5-point Likert scale with the following score definitions, depending on the question: 0 = not at all (or none of the time), 1 = a little bit (or a little of the time), 2 = moderately (or some of the time), 3 = quite a bit (or most of the time), and 4 = extremely (or all of the time). The total score is the mean of all non-missing items. The range of the total score is 0 (response is 'not at all' for each item) to 4 (response is 'extremely' for each item). Negative change from baseline values indicate improvement in constipation quality of life. Each participant completed the PAC-QOL at Baseline and Week 52 using a 2-week recall period.
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PAC-QOL data. Two participants were randomized to the Placebo Arm but were administered CB-5945 instead. As a result, these 2 participants were included in the CB-5945 Arm for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CB-5945 | Placebo
Number analyzed (Participants) | 240 | 236
units on a scale | -0.63 (0.699) | -0.45 (0.583)

4. Secondary Outcome: Change From Baseline in Patient-Reported Constipation Severity Assessment (PCSA) at Week 52
Description: The PCSA asked participants to rate the severity of their overall constipation during the 24 hours prior to the assessment, using a scale of 0 to 10, where 0 is no constipation and 10 is the worst constipation imaginable.
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PCSA data. Two participants were randomized to the Placebo Arm but were administered CB-5945 instead. As a result, these 2 participants were included in the CB-5945 Arm for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CB-5945 | Placebo
Number analyzed (Participants) | 208 | 193
units on a scale | -3.0 (3.24) | -2.2 (3.19)

5. Secondary Outcome: Plasma Trough Concentrations of CB-5945
Description: Blood samples for trough concentrations of CB-5945 were collected before the participant's morning dose of study drug at Weeks 4, 12, 24, 36, and 52. Overall concentration was based on the mean trough level for each participant across all weeks.
Time Frame: Weeks 4, 12, 24, 36, and 52
Population: All participants randomized to CB-5945 who received at least 1 dose of study drug and had evaluable CB-5945 concentration data. Two participants were randomized to the Placebo Arm but were administered CB-5945 instead. As a result, these 2 participants were included in the CB-5945 Arm for analysis.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | CB-5945
Number analyzed (Participants) | 631
picograms per milliliter (pg/mL)
  Week 4 (n=615) | 517.51 (403.391)
  Week 12 (n=522) | 549.66 (425.131)
  Week 24 (n=419) | 547.31 (453.548)
  Week 36 (n=288) | 573.57 (517.118)
  Week 52 (n=203) | 616.57 (725.849)
  Overall (n=631) | 517.19 (375.963)

6. Other Pre Specified Outcome: Number of Participants With Adjudicated Cardiovascular, Gastrointestinal, or Central Opioid Withdrawal Events
Description: Cardiovascular (CV) events of interested included mycardial infarction, unstable angina, CV accident, congestive heart failure, serious arrhythmia, resuscitated cardiac arrest, and death.
  Gastrointestinal (GI) events of interest included emergency department visits for the serious adverse events of gastroenteritis, hepatitis, pancreatitis, nausea, vomiting, diarrhea, and abdominal pain or cramping.
  Central opioid withdrawal (OW) events of interest included opioid withdrawal syndrome. The adverse events that indicated central OW included, but were not limited to, hyperhidrosis, tremor, dysphoria, and myalgia.
  The number of participants with at least 1 confirmed CV, GI, or Central OW event is presented.
Time Frame: Baseline through Week 56
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | CB-5945 | Placebo
Number analyzed (Participants) | 703 | 700
participants
  CV event | 1 | 2
  GI event | 16 | 7
  Central OW event | 7 | 2

ADVERSE EVENTS:
Description: Two participants were randomized to the Placebo Arm but were administered CB-5945 instead. As a result, these 2 participants were included in the CB-5945 Arm for analysis.
Arm/Group | CB-5945 | Placebo
Serious Adverse Events (participants affected / at risk) | 40/703 | 36/700
Other Adverse Events (participants affected / at risk) | 403/703 | 373/700
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | CB-5945 (N=703) | Placebo (N=700)
Gastroenteritis (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 1 | 3
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Infected bites (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Meningitis staphylococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Faecaloma (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/437 | 0/417
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/437 | 1/417
Psychotic disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1
Violence-related symptom (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | CB-5945 (N=703) | Placebo (N=700)
Diarrhoea (Gastrointestinal disorders) | 90 | 33
Abdominal Pain (Gastrointestinal disorders) | 57 | 32
Nausea (Gastrointestinal disorders) | 51 | 39
Vomiting (Gastrointestinal disorders) | 35 | 20
Abdominal Pain Upper (Gastrointestinal disorders) | 20 | 11
Flatulence (Gastrointestinal disorders) | 17 | 16
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 9 | 2
Constipation (Gastrointestinal disorders) | 8 | 11
Abdominal Distension (Gastrointestinal disorders) | 7 | 8
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Haemorrhoids (Gastrointestinal disorders) | 4 | 6
Abdominal Discomfort (Gastrointestinal disorders) | 3 | 4
Abdominal Pain Lower (Gastrointestinal disorders) | 3 | 2
Haematochezia (Gastrointestinal disorders) | 3 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 3 | 3
Colonic Polyp (Gastrointestinal disorders) | 2 | 1
Faecal Incontinence (Gastrointestinal disorders) | 2 | 2
Frequent Bowel Movements (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Abdominal Tenderness (Gastrointestinal disorders) | 1 | 0
Abdominal Wall Mass (Gastrointestinal disorders) | 1 | 0
Anorectal Discomfort (Gastrointestinal disorders) | 1 | 0
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Bowel Movement Irregularity (Gastrointestinal disorders) | 1 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 3
Dry Mouth (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Erosive Oesophagitis (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 1
Faeces Discoloured (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastric Polyps (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gingival Pain (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 2
Oral Papule (Gastrointestinal disorders) | 1 | 0
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0
Rectal Discharge (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 0
Abdominal Adhesions (Gastrointestinal disorders) | 0 | 1
Abnormal Faeces (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Rectal Spasm (Gastrointestinal disorders) | 0 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 3
Urinary Tract Infection (Infections and infestations) | 25 | 22
Upper Respiratory Tract Infection (Infections and infestations) | 18 | 28
Bronchitis (Infections and infestations) | 17 | 10
Nasopharyngitis (Infections and infestations) | 17 | 13
Sinusitis (Infections and infestations) | 17 | 22
Gastroenteritis Viral (Infections and infestations) | 16 | 12
Influenza (Infections and infestations) | 13 | 12
Gastroenteritis (Infections and infestations) | 8 | 5
Tooth Abscess (Infections and infestations) | 8 | 7
Pneumonia (Infections and infestations) | 6 | 6
Ear Infection (Infections and infestations) | 4 | 2
Oral Candidiasis (Infections and infestations) | 4 | 0
Laryngitis (Infections and infestations) | 3 | 0
Pharyngitis Streptococcal (Infections and infestations) | 3 | 2
Atypical Pneumonia (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 2
Eye Infection (Infections and infestations) | 2 | 0
Furuncle (Infections and infestations) | 2 | 1
Localised Infection (Infections and infestations) | 2 | 3
Staphylococcal Infection (Infections and infestations) | 2 | 1
Tooth Infection (Infections and infestations) | 2 | 4
Viral Infection (Infections and infestations) | 2 | 2
Vulvovaginal Mycotic Infection (Infections and infestations) | 2/437 | 0/417
Bacteriuria (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis Of Male External Genital Organ (Infections and infestations) | 1/266 | 0/283
Chronic Sinusitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 3
Ear Infection Bacterial (Infections and infestations) | 1 | 0
Gastritis Viral (Infections and infestations) | 1 | 1
Gastrointestinal Viral Infection (Infections and infestations) | 1 | 0
Herpes Dermatitis (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 2
Impetigo (Infections and infestations) | 1 | 0
Infected Bites (Infections and infestations) | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 1
Otitis Media (Infections and infestations) | 1 | 1
Papilloma Viral Infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 3
Pyelonephritis (Infections and infestations) | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Sinusitis Bacterial (Infections and infestations) | 1 | 0
Staphylococcal Skin Infection (Infections and infestations) | 1 | 0
Vaginitis Bacterial (Infections and infestations) | 1/437 | 1/417
Viral Diarrhoea (Infections and infestations) | 1 | 0
Acute Sinusitis (Infections and infestations) | 0 | 2
Chlamydial Infection (Infections and infestations) | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 2
Gastroenteritis Norovirus (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Genital Herpes (Infections and infestations) | 0 | 1
Herpes Simplex (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 2
Oesophageal Candidiasis (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Skin Candida (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 2
Tinea Pedis (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 31 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 14
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 10 | 11
Neck Pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8 | 11
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 7
Joint Swelling (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 3 | 3
Foot Deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 | 3
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 20 | 23
Neuralgia (Nervous system disorders) | 8 | 5
Dizziness (Nervous system disorders) | 5 | 10
Hypoaesthesia (Nervous system disorders) | 4 | 0
Migraine (Nervous system disorders) | 4 | 5
Sinus Headache (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 3 | 2
Dysgeusia (Nervous system disorders) | 2 | 1
Neuropathy Peripheral (Nervous system disorders) | 2 | 5
Restless Legs Syndrome (Nervous system disorders) | 2 | 1
Sciatica (Nervous system disorders) | 2 | 2
Somnolence (Nervous system disorders) | 2 | 0
Tension Headache (Nervous system disorders) | 2 | 0
Amnesia (Nervous system disorders) | 1 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 5
Complex Regional Pain Syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Diabetic Neuropathy (Nervous system disorders) | 1 | 0
Drooling (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Migraine With Aura (Nervous system disorders) | 1 | 0
Mononeuropathy (Nervous system disorders) | 1 | 0
Narcolepsy (Nervous system disorders) | 1 | 1
Occipital Neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Parkinson's Disease (Nervous system disorders) | 1 | 0
Peroneal Nerve Palsy (Nervous system disorders) | 1 | 0
Speech Disorder (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 3
Cognitive Disorder (Nervous system disorders) | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 0 | 1
Muscle Contractions Involuntary (Nervous system disorders) | 0 | 1
Radiculitis (Nervous system disorders) | 0 | 1
Tarsal Tunnel Syndrome (Nervous system disorders) | 0 | 1
Drug Withdrawal Syndrome (General disorders) | 10 | 7
Pain (General disorders) | 9 | 4
Fatigue (General disorders) | 8 | 6
Oedema Peripheral (General disorders) | 4 | 13
Pyrexia (General disorders) | 4 | 3
Chest Discomfort (General disorders) | 2 | 0
Chest Pain (General disorders) | 2 | 0
Chills (General disorders) | 2 | 1
Influenza Like Illness (General disorders) | 2 | 3
Medical Device Pain (General disorders) | 2 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 2
Oedema (General disorders) | 2 | 3
Adverse Drug Reaction (General disorders) | 1 | 1
Feeling Cold (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Spinal Pain (General disorders) | 1 | 0
Temperature Intolerance (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Face Oedema (General disorders) | 0 | 1
Tenderness (General disorders) | 0 | 1
Ulcer (General disorders) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 5 | 5
Muscle Strain (Injury, poisoning and procedural complications) | 5 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 4 | 1
Excoriation (Injury, poisoning and procedural complications) | 4 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 4
Foot Fracture (Injury, poisoning and procedural complications) | 4 | 2
Laceration (Injury, poisoning and procedural complications) | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 7
Head Injury (Injury, poisoning and procedural complications) | 2 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 2 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 2
Tendon Rupture (Injury, poisoning and procedural complications) | 2 | 0
Accidental Exposure (Injury, poisoning and procedural complications) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 2
Heat Exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 1
Lip Injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 3
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 1
Suture Rupture (Injury, poisoning and procedural complications) | 1 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 1
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 | 2
Anal Injury (Injury, poisoning and procedural complications) | 0 | 1
Burns Second Degree (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 0 | 3
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Allergic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Hyperinflation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis Seasonal (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 10 | 4
Insomnia (Psychiatric disorders) | 7 | 9
Depression (Psychiatric disorders) | 6 | 9
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 3 | 2
Confusional State (Psychiatric disorders) | 2 | 0
Mood Swings (Psychiatric disorders) | 2 | 0
Restlessness (Psychiatric disorders) | 2 | 1
Affective Disorder (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 1 | 3
Generalised Anxiety Disorder (Psychiatric disorders) | 0 | 1
Initial Insomnia (Psychiatric disorders) | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 2
Panic Attack (Psychiatric disorders) | 0 | 1
Sleep Disorder (Psychiatric disorders) | 0 | 2
Tobacco Withdrawal Symptoms (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 14 | 8
Hot Flush (Vascular disorders) | 8 | 6
Hypotension (Vascular disorders) | 4 | 4
Raynaud's Phenomenon (Vascular disorders) | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1
Peripheral Vascular Disorder (Vascular disorders) | 0 | 1
Post Thrombotic Syndrome (Vascular disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 5
Cold Sweat (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 6
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Increased Tendency To Bruise (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 2
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Piloerection (Skin and subcutaneous tissue disorders) | 1 | 1
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 3
Alanine Aminotransferase Increased (Investigations) | 4 | 0
Weight Increased (Investigations) | 4 | 2
Aspartate Aminotransferase Increased (Investigations) | 3 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 2 | 2
Blood Lactate Dehydrogenase Increased (Investigations) | 2 | 0
Blood Pressure Increased (Investigations) | 2 | 2
Blood Uric Acid Increased (Investigations) | 2 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 2 | 2
Haemoglobin Decreased (Investigations) | 2 | 0
Hepatic Enzyme Increased (Investigations) | 2 | 3
Neutrophil Count Increased (Investigations) | 2 | 0
Platelet Count Increased (Investigations) | 2 | 0
Aortic Bruit (Investigations) | 1 | 0
Blood Cholesterol Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 1
Blood Glucose Increased (Investigations) | 1 | 0
Blood Sodium Increased (Investigations) | 1 | 0
Blood Triglycerides Increased (Investigations) | 1 | 1
Glomerular Filtration Rate Increased (Investigations) | 1 | 0
Haematocrit Decreased (Investigations) | 1 | 0
Heart Rate Increased (Investigations) | 1 | 0
Liver Function Test Abnormal (Investigations) | 1 | 2
Monocyte Count Decreased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0
Red Blood Cell Count Decreased (Investigations) | 1 | 0
Urine Phosphorus Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 1 | 1
White Blood Cell Count Increased (Investigations) | 1 | 3
Blood Phosphorus Decreased (Investigations) | 0 | 1
Blood Sodium Decreased (Investigations) | 0 | 1
Blood Testosterone Decreased (Investigations) | 0 | 1
Blood Urine Present (Investigations) | 0 | 1
Cardiac Murmur (Investigations) | 0 | 1
Crystal Urine Present (Investigations) | 0 | 1
Electrocardiogram Qt Prolonged (Investigations) | 0 | 1
Fungal Test Positive (Investigations) | 0 | 1
Glomerular Filtration Rate Decreased (Investigations) | 0 | 1
Haematocrit Increased (Investigations) | 0 | 1
Heart Rate Decreased (Investigations) | 0 | 1
Transaminases Increased (Investigations) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 7
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 4
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 7 | 6
Haematuria (Renal and urinary disorders) | 3 | 3
Chromaturia (Renal and urinary disorders) | 1 | 0
Diabetic Nephropathy (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 2
Glycosuria (Renal and urinary disorders) | 1 | 0
Hypertonic Bladder (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 2
Renal Impairment (Renal and urinary disorders) | 1 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Renal Injury (Renal and urinary disorders) | 0 | 1
Lacrimation Increased (Eye disorders) | 4 | 2
Cataract (Eye disorders) | 3 | 2
Conjunctivitis (Eye disorders) | 2 | 3
Blepharitis (Eye disorders) | 1 | 0
Blindness Unilateral (Eye disorders) | 1 | 0
Dry Eye (Eye disorders) | 1 | 0
Eye Pruritus (Eye disorders) | 1 | 1
Eyelid Ptosis (Eye disorders) | 1 | 1
Panophthalmitis (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 1 | 1
Conjunctival Haemorrhage (Eye disorders) | 0 | 1
Iritis (Eye disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 2
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus Arrhythmia (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 2
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 2/437 | 0/417
Breast Disorder (Reproductive system and breast disorders) | 1 | 1
Breast Mass (Reproductive system and breast disorders) | 1 | 1
Breast Pain (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1/437 | 0/417
Genital Rash (Reproductive system and breast disorders) | 1 | 0
Vaginal Lesion (Reproductive system and breast disorders) | 1/437 | 0/417
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0/266 | 1/283
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0/437 | 1/417
Erectile Dysfunction (Reproductive system and breast disorders) | 0/266 | 1/283
Prostatomegaly (Reproductive system and breast disorders) | 0/266 | 1/283
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0/437 | 1/417
Anaemia (Blood and lymphatic system disorders) | 5 | 7
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Cyst (Hepatobiliary disorders) | 1 | 0
Hepatic Mass (Hepatobiliary disorders) | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 1 | 0
Liver Disorder (Hepatobiliary disorders) | 1 | 0
Biliary Dilatation (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Seasonal Allergy (Immune system disorders) | 2 | 3
Allergy To Arthropod Bite (Immune system disorders) | 1 | 0
Allergy To Metals (Immune system disorders) | 1 | 0
Allergy To Vaccine (Immune system disorders) | 0 | 1
Cerumen Impaction (Ear and labyrinth disorders) | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2
Goitre (Endocrine disorders) | 1 | 0
Hypogonadism (Endocrine disorders) | 1 | 1
Adrenal Mass (Endocrine disorders) | 0 | 1
Androgen Deficiency (Endocrine disorders) | 0 | 1
Hypogonadism Male (Endocrine disorders) | 0/266 | 1/283
Hypothyroidism (Endocrine disorders) | 0 | 3
Tooth Extraction (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other